CLINICAL TRIAL: NCT07206875
Title: Retrospective and Prospective Observational Registry for the Characterisation of Patients Affected by Any Type of Diabetes and Endocrine-metabolic Disorders
Brief Title: Observational Study for the Characterisation of Patients Affected by Any Type of Diabetes and Endocrine Disorders
Acronym: DiabRegistry
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, EMANUELA SETOLA, MEDICAL DOCTOR, IRCCS San Raffaele
Other Study IDs: DiabRegistry
Record Dates: First submitted 2025-07-23; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Diabetes; Metabolic Disorders; Arterial Hypertension; Dyslipidemia; Liver Disease (Alcoholic or Not)
Keywords: diebetes; metabolic disorders; endocrine disorders; observational study
MeSH Terms: conditions — Diabetes Mellitus; Metabolic Diseases; Hypertension; Dyslipidemias; Liver Diseases; Endocrine System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Endocrine-metabolic-disase participants

SUMMARY:
The main objective of this retrospective and prospective observational register is to identify anthropometric, clinical, laboratory and/or instrumental markers of disease severity and activity in patients suffering from diabetes, endocrine-metabolic disorders, rare diseases in order to improve their diagnosis, monitoring and treatment processes. The Registry is monocentric, observational prospective and retrospective. No additional procedures to those of normal clinical practice are planned, and neither diagnostic approaches nor experimental drugs/prescriptions will be applied. The data under study (demographic, anthropometric, clinical and care characteristics) will be collected as part of outpatient visits of the Diabetes Outpatient Clinic or admission to Diabetes Day Hospital.

In case of outpatients, the observation will start at the diagnosis or during the first outpatient visit and will end with the last outpatient visit performed within the total time foreseen for the duration of the study.

The study will start once the regulatory authorizations are completed, and is expected to last at least 10 years with the possibility of extension

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Outpatient Diabetes Unit patient
* Ability to give informed consent

Diagnosis of at least one of the following:

* Metabolic disease, defined as BMI ≥25 Kg/m2
* Type 1 or type 2 diabetes mellitus
* Gestational diabetes
* Monogenic diabetes (MODY)
* Other types of diabetes or dysglycemia
* Dyslipidemia
* Arterial hypertension
* Steatosis liver disease (SLD)

Exclusion Criteria:

* Age <18 years
* Deny participation at the study
* Recruitment in an interventional protocol
* Patients with missing significant data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diabetes and endocrine-metabolic diseases accessing the care services of the O.U. of Diabetology
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2035-11 (Estimated)

PRIMARY OUTCOMES:
GLUCOSE | baseline
  glucose in milligrams per deciliter;
HBA1C | baseline
  glycates hemoglobin in millimoles per mole.
Insulin | baseline
  insulin in microunits per milliliter;
UACR | baseline
  Urine analysis: albumine in milligrams per liter, creatinine millimoles per liter.
Anthropometric parameters | baseline
  BMI: body mass index : weight/height2 = kilogram/cm2
c-pep | baseline
  c-peptide in nanograms per milliliter;

CONTACTS AND LOCATIONS:
Locations (1):
- Diabetology Department, San Raffaele Scientific Institute, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: Undecided